CLINICAL TRIAL: NCT03933865
Title: Acute Pain Management in Patients on Opioid Replacement Therapy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The COVID-19 pandemic and recruitment difficulties prompted the investigators to terminate study early.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Z-1701
Record Dates: First submitted 2018-12-04; First posted 2019-05-01 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Opioid-use Disorder; Pain, Acute
Keywords: buprenorphine; quantitative sensory testing; cold pressor; abuse liability; ketamine; hydromorphone
MeSH Terms: conditions — Opioid-Related Disorders; Acute Pain | interventions — Hydromorphone; Ketamine

STUDY DESIGN:
Intervention Model Description: This is an outpatient randomized within subject placebo-controlled human laboratory investigation of analgesia (as assessed with quantitative sensory testing) from ketamine alone and in combination with hydromorphone in buprenorphine maintained participants.
Masking Description: Masking: Participant, Investigator, and Outcomes Assessor. The identity of study medication conditions will not be known to investigators, research staff, or patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Buprenorphine Maintained Patients (Other): All participants will be maintained on buprenoprhine for the treatment of opioid use disorder. All participants will be exposed to all 8 study drug combinations
  Interventions: Drug: HYDROmorphone Injectable Solution; Drug: Ketamine; Drug: Placebos

INTERVENTIONS:
Drug: HYDROmorphone Injectable Solution — Hydromorphone will be given via intramuscular injection (8 mg)
  Other Names: Dilaudid
Drug: Ketamine — Ketamine will be given via intramuscular injection (0.1, 0.2 or 0.4 mg/kg)
Drug: Placebos — Placebo will be normal saline solution given via intramuscular injection.

SUMMARY:
This is an outpatient randomized within subject placebo-controlled human laboratory investigation of analgesia (as assessed with quantitative sensory testing; QST) from ketamine alone and in combination with hydromorphone in buprenorphine maintained participants. The goals of this project are to characterize the analgesic, subjective, and physiologic effects of ketamine combined with hydromorphone in patients on buprenorphine maintenance for opioid use disorder.

DETAILED DESCRIPTION:
Eligible participants will have 8 sessions where they will receive two IM injections.The dose of ketamine will be manipulated (0 mg/kg to 0.4 mg/kg) across sessions. The dose of hydromorphone will either be 0 mg or 8 mg. Therefore, participants will be exposed to ascending doses of ketamine with and without hydromorphone. Order of study medications will be randomized for each participant by an un-blinded statistician and transmitted securely to study pharmacist in charge of medication administration. This study will provide unique information on optimal hydromorphone-ketamine dosing strategies for acute pain management. in buprenorphine maintained patients.

Each session will take place 17 hours after the last buprenorphine dose (trough levels) to control for time since last dose. Sessions will be held on a dedicated unit for human subjects clinical research at Zuckerberg San Francisco General and include two IM injections of study medication given 15 minutes apart by blinded nursing staff. Study sessions will each last approximately 5 hours. Sessions will take place 1-2x weekly and must be separated by at least 72 hours to allow for drug wash-out. QST outcomes will be measured at baseline, as well as 15, 75, 135, and 195 minutes after injection #2 for each session. In addition, abuse liability outcomes will be measured at baseline (if required) and at 15, 75, 135, and 195 minutes after injection #2 for each session.

Blood will be drawn to evaluate baseline buprenorphine /norbuprenorphine levels. Then, PK analyses will be done for ketamine, norketamine and hydromorphone. Blood will be drawn at baseline as well as 15, 75, 135, and 195 minutes after injection #2.

Primary outcome will be analgesia as assessed by QST. The use of various QST measures which assess acute anti-nociception as well as central modification of pain processing will allow us to evaluate whether overall analgesia results from blocking of nociceptor signaling and/or changes to central pain facilitation to better understand the mechanism of ketamine-hydromorphone combinations.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 18-60 years of age, inclusive.
2. Maintained on stable buprenorphine/naloxone (Suboxone®) dose for at least 30 days prior to screening, with total daily dose >=4 mg and <=24 mg (Patients may also be on Zubsolv ® equivalent doses >=2.9 and <=17.2 mg). Participant must agree to stay on this dose for duration of study participation.
3. Urine toxicology screen negative for drugs of abuse but positive for buprenorphine.
4. Willing and able to speak, read and understand English.
5. Able and willing to perform/tolerate QST. Persons who can tolerate cold pressor testing for 5 minutes will be disqualified.
6. Willing to abstain from analgesic medications (other than buprenorphine) for 24 hours prior to each session.
7. Written informed consent obtained from participant and ability for participant to comply with the requirements of the study.

Exclusion Criteria:

1. Current alcohol or sedative-hypnotic use disorder as assessed by the Mini International Neuropsychiatric Interview.
2. Presence of acute or chronic pain as determined by medical history and physical examination and score of 0 on pain VAS at the start of experimental sessions.
3. Medical or psychiatric condition known to influence QST (e.g. HIV, peripheral neuropathy, Schizophrenia, Raynaud's syndrome).
4. Women who are pregnant, breastfeeding, or planning on becoming pregnant during course of trial. Women must be using effective birth control and will receive pregnancy tests before each session.
5. Poor venous access as an IV catheter will be used for blood draws during sessions.
6. Past history of psychotic disorder (as assessed through MINI).
7. Uncontrolled hypertension or clinically significant ECG abnormality.
8. History of allergy or significant adverse reaction to hydromorphone or ketamine.
9. Significant contraindication to ketamine use (active psychosis, uncontrolled hypertension, past or current ketamine use disorder, cardiovascular disease, glaucoma, active pulmonary infection or disease).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2022-02-24 (Actual); Study Completion 2022-02-24 (Actual)

PRIMARY OUTCOMES:
peak change in cold pressor tolerance | 1 day per session
  The amount of time (seconds) a participant can keep hand in cold water bath before pain becomes unbearable. The change will be the highest value after study medications have been administered subtracted from the session baseline.

SECONDARY OUTCOMES:
peak change in cold pressor threshold | 1 day per session
  The time (seconds) at which pain first develops after placing hand in cold water bath. The change will be the highest value after study medications have been administered subtracted from the session baseline.
peak change in conditioned pain modulation (CPM) | 1 day per session
  Responses to a brief pressure pain stimulus are evaluated alone and then re-assessed during application of a tonic noxious stimulus (hand in water bath) using validated procedures. The peak change in CPM outcome will be a difference in differences score: the largest value of CPM after study medications have been administered subtracted from CPM at baseline

OTHER OUTCOMES:
Peak Drug Liking Visual Analog Scale | 1 day per session
  The participant positions an arrow along a line (labeled from 0 to 100) using the keypad to indicate his or her answer of how s/he likes the drug(s) at that moment.

CONTACTS AND LOCATIONS:
Overall Officials: D. Andrew Tompkins, MD MHS, Principal Investigator — University of California, San Francisco
Locations (1):
- Zuckerberg San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No